## **CCB-CRISIS-01**

# THE CRISIS STUDY: A RANDOMIZED OPEN-LABEL STUDY ASSESSING THE SAFETY AND ANTI-CORONAVIRUS RESPONSE OF SUPPRESSION OF HOST NUCLEOTIDE SYNTHESIS IN HOSPITALIZED ADULTS WITH CORONAVIRUS-19 (COVID-19)

## NCT04425252

STATISTICAL ANALYSIS PLAN DATE: 17-DEC-2020



## Statistical Analysis Plan

| Sponsor: | Clear Creek Bio, Inc |
|---|---|
| Protocol No: | CCB-CRISIS-01 |
| Protocol Title: | A randomized open-label study assessing the safety and anti-coronavirus response of suppression of host nucleotide synthesis in hospitalized adults with coronavirus-19 (COVID-19) |
| Document Date: | 17-Dec-2020 |
| Document Revision | 1.0 |

Doc. No.: TMP-BS-01

Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


## **APPROVAL SIGNATURES**

#### Prosoft Personnel

| Title | Printed Name | Signature | Date |
|---|---|---|---|
| Manager,<br>Statistics | Daisy Chen | DocuSigned by: Daisy (lun Signer Name: Daisy Chen | 17-Dec-2020 |
| Associate Vice<br>President, Statistics | Diane Tipping | Signing Reason: I have reviewed this do<br>Signing Time: 17-Dec-2020 1:30:14 PN<br>2B3FFE99115C431EB126300C7C7DA | |
| CCD D | | Signer Name: Diane Tipping Signing Reason: I approve this docume Signing Time: 17-Dec-2020 4:32:51 P | M EST |

#### **CCB Personnel**

| Title | Printed Name | Signature | Date |
|---|---|---|---|
| Vice President,<br>Clinical Operations | Barbara Powers, PhD | DocuSigned by: Barbara Powers Signer Name: Barbara Powers | 17-Dec-2020 |
| | | Signing Reason: I approve this document Signing Time: 17-Dec-2020 1:39:56 PM PST | |

-57DEAAD17C2240FEA72C57ABA124E827

## **DOCUMENT HISTORY**

| Rev No | Date | Description |
|--------|-------------|-------------------|
| 1.0 | 17-Dec-2020 | Original document |

#### Confidential Document

Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


## TABLE OF CONTENTS

| 1. | INT | FRODUCTION | | 6 |
|----|------|--------------------|--------------------------------|----|
| | 1.1 | Background | | 6 |
| | 1.2 | Trial Design | | 6 |
| | 1.2. | 1 Number of Sul | ubjects and Randomization | 7 |
| | 1.3 | Trial Objectives | | 7 |
| | 1.3. | 1 Primary Object | ctives | 7 |
| | 1.3. | 2 Secondary Obj | pjectives | 7 |
| | 1.3. | 3 Exploratory O | Objectives | 7 |
| 2. | ST | ATISTICAL MET | THODOLOGY | 7 |
| | 2.1 | General Principles | S | 7 |
| | 2.2 | Sample Size Determ | mination | 8 |
| | 2.3 | Trial Populations | | 8 |
| | 2.4 | Subject Accounting | g and Baseline Characteristics | 8 |
| | 2.5 | Efficacy Analyses. | | 8 |
| | 2.5. | 1 Primary Effica | acy Analyses | 8 |
| | 2.5. | 2 Secondary Eff | ficacy Analyses | 8 |
| | 2.5. | 3 Exploratory E | Efficacy Analyses | 9 |
| | 2.6 | Safety Analyses | | 10 |
| | 2.7 | Interim Analyses | | 11 |
| 3. | DA | TA HANDLING | | 11 |
| | 3.1 | Baseline and Study | y Visits | 11 |

Doc No.: TMP-BS-01

Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020 

| | NDIX 1 CTCAE V4 03 GRADING FOR LABORATORY VALUES | |
|-------|--------------------------------------------------|----|
| 4. CF | HANGES FROM THE PROTOCOL | 14 |
| 3.3 | Missing Data and Data Conventions | 13 |
| 3.2 | Derived Data | 11 |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


## List of Abbreviations

| AE | Adverse Event |
|------------|-------------------------------------------------|
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| CI | Confidence Interval |
| COVID-19 | Coronavirus Disease 2019 |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DHO | Dihydroorotate |
| DHODH | Dihydroorotate Dehydrogenase |
| DSMB | Data Safety Monitoring Board |
| EHR | Electronic Health Record |
| ICU | Intensive Care Unit |
| LLN | Lower Limit of Normal |
| LLOQ | Lower Limit of Quantification |
| mITT | Modified Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NEWS2 | National Early Warning System 2 |
| Q1 | First Quartile |
| Q3 | Third Quartile |
| RNA | Ribonucleic Acid |
| SARS-CoV-2 | Severe Acute Respiratory Syndrome Coronavirus 2 |
| SE | Standard Error |
| SOC | Standard of Care |
| TEAE | Treatment-Emergent Adverse Event |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cell |
| WHODrug | World Health Organization Drug Dictionary |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


#### 1. INTRODUCTION

### 1.1 Background

Beginning in December 2019, Chinese scientists isolated a novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) from patients with virus-infected pneumonia which was later designated as coronavirus disease 2019 (COVID-19) by the World Health Organization (WHO). Approximately 14% of those affected with this virus will develop severe disease requiring hospitalization and oxygen support; 5% will require admission to the intensive care unit (ICU). Coronaviruses, like other Ribonucleic acid (RNA) based viruses, do not have the machinery to synthesize their own nucleotides and thus depend upon the host intracellular pool of nucleotides for viral replication. In essence, viruses steal the host RNA building blocks, and without these building blocks they are unable to replicate.

Dihydroorotate dehydrogenase (DHODH) is a clear therapeutic target for the inhibition of host pyrimidine synthesis. Brequinar is an orally available and potent inhibitor of DHODH. Brequinar is one of more than 300 quinoline-carboxylic acid derivatives prepared in an analog synthesis program in the 1980s, which was started after it was found that a compound of this class had antitumor activity.

The CRISIS trial will study standard of care (SOC) and SOC with 5 days of DHODH inhibition. Clear Creek Bio hypothesizes that a defined 5-day course of brequinar will inhibit the enzyme DHODH to a degree sufficient to result in the transient depletion of host pyrimidine nucleotides, thereby inhibiting viral replication.

## 1.2 Trial Design

This will be a phase 1a randomized, open label, multi-center study with approximately 24 subjects. All subjects will receive SOC per institutional guidelines for treatment of patients with COVID-19 infection. In addition to SOC, the brequinar group will receive brequinar 100 mg once daily for 5 days.

Subjects will have a Screening Visit followed as soon as possible with Study Day 1 (Day 1 may take place on the same day if entry criteria data are available). Subjects will be followed through Day 15, with mortality assessed via a phone call/other digital media acceptable to institution on Day 29.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


## 1.2.1 Number of Subjects and Randomization

Subjects who meet all the inclusion and none of the exclusion criteria will be enrolled in the study until approximately 24 subjects have completed the study. Subjects will be randomized to either SOC or SOC plus brequinar or in a 1:2: ratio (approximately 8 subjects assigned to SOC alone and approximately 16 subjects on SOC plus brequinar).

## 1.3 Trial Objectives

## 1.3.1 Primary Objectives

The primary objective of this study is to determine the safety and tolerability of SOC and SOC plus brequinar in hospitalized COVID-19 subjects.

## 1.3.2 Secondary Objectives

The secondary objectives of this study are

- To determine the changes in clinical status measures through Day 15
  - o hospitalization status
  - o duration of hospitalization
  - o NEWS2 Score
- To determine survival status through Day 29

## 1.3.3 Exploratory Objectives

- To determine the change in SARS-CoV-2 nasopharyngeal viral load through Day 15
- To determine the change in inflammatory markers through Day 15
- To determine the change in DHO levels through Day 15
- To determine the change in brequinar concentration levels through Day 7

#### 2. STATISTICAL METHODOLOGY

## 2.1 General Principles

In general, continuous parameters will be summarized by number of non-missing observations (N), mean, standard error (SE), median, quartiles, minimum, and maximum. Categorical parameters will be summarized by count and percentage of the non-missing observations, and


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


95% confidence interval (CI), when appropriate. All statistical analyses will be performed using SAS® Version 9.4. Adverse events (AEs), procedures and medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 23.0. Prior and concomitant medications will be coded using World Health Organization Drug Dictionary (WHODrug) Enhanced March 2020. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 will be utilized for adverse event and laboratory reporting.

All study data collected will be presented in listings.

## 2.2 Sample Size Determination

Formal sample size calculations are not applicable for this phase 1a, open label study. Up to 24 subjects are planned to be entered in this trial. Additional subjects may be enrolled following data review.

### 2.3 Trial Populations

The modified Intent to Treat (mITT) population will include all randomized subjects who had at least one post-randomization assessment, and who received at least one dose of study medication if randomized to SOC + Brequinar group. All analyses will be based on the mITT population.

## 2.4 Subject Accounting and Baseline Characteristics

Demographics and baseline characteristics (including NEWS2 score and ICU level of care at randomization) will be summarized by treatment. Prior and concomitant medications/procedures will be summarized by treatment. A medication/procedure may be classified as both prior and concomitant. Medical history will be summarized by treatment.

## 2.5 Efficacy Analyses

## 2.5.1 Primary Efficacy Analyses

None

## 2.5.2 Secondary Efficacy Analyses

#### **Hospitalization Status and Duration**

Hospitalization status (died, hospitalized in ICU, hospitalized not in ICU, discharged for initial hospitalization and re-hospitalization) will be summarized on Study Day 3, 5, 7 and 15. Kaplan Confidential Document

Doc No.: TMP-BS-01

Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


Meier estimates and plots will be provided to assess the duration of hospitalization (Study Day at time of initial discharge). Subjects who were not discharged by the Day 15 visit will be censored at the Day 15 visit. Subjects who did not complete the trial while still hospitalized will be censored at the date of last contact.

#### **NEWS2 Score**

Changes from baseline to Day 3, 5, 7, and 15 in NEWS2 scores will be summarized by treatment. In addition, the NEWS2 scores will be summarized by category (0-4, 5-6, 7 or above). The NEWS2 parameters will be summarized at each visit, including changes from baseline for continuous parameters. (See Section 3.2 for derivation of NEWS2 score).

#### Mortality

Mortality will be summarized through Day 29 by treatment group. Kaplan Meier estimates and plots will be provided to assess the time to death (date of death minus date of randomization). Subjects who are alive at the Day 29 contact will be censored at the Day 29 contact. Subjects whose Day 29 survival is unknown will be censored at the date of last contact.

## 2.5.3 Exploratory Efficacy Analyses

Changes from baseline will be summarized by treatment:

- Viral load (nasopharyngeal) (Days 3, 5, 7, and 15)
- Inflammatory markers (Days 3, 5, 7, and 15)
- DHO levels (Days 3, 5, 7, and 15)
- Brequinar concentration levels (Days 3, 5 and 7)

For inflammatory markers (including pro-inflammatory cytokines), results from both local and central laboratories will be combined, where the local test result will be normalized where necessary. (See Section 3.2 for normalization method).

Viral culture results will be provided in data listings only.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


#### 2.6 Safety Analyses

#### **Adverse Events**

An overall summary of treatment-emergent adverse events (TEAEs) will be presented by treatment and total, including the total number of events, frequency counts and percentages for:

- o Any TEAE
- o Treatment-related TEAEs
- CTCAE Grade 3 or above TEAEs
- TEAEs leading to drug withdrawn
- o TEAEs leading to study discontinuation
- Serious TEAEs
- o Fatal TEAEs
- o TEAEs of interest

The incidence of TEAEs by treatment and total will be tabulated by MedDRA system organ class and preferred term for:

- o All TEAEs
- o Treatment-related TEAEs
- o TEAEs by severity
- o TEAEs leading to study discontinuation
- Serious TEAEs
- o TEAEs of interest

AEs will be considered treatment-emergent if the onset date is on or after the day of randomization. "Drug related" will include 'Definite', 'Probable' and 'Possible' relationship to drug as determined by the Investigator.

#### **Safety Laboratory Assessments**

Safety laboratory tests (Chemistry and Hematology) will be performed throughout the study. Laboratory parameters of interest (AST, ALT, ALP, Total Bilirubin, Creatinine, Hemoglobin, WBC, Absolute Neutrophils, Absolute Lymphocytes and Platelets) will be summarized for changes from baseline.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


NCI CTCAE grades will be derived for the lab parameters included in Appendix 1 and presented in data listings. Separate listings of Grade 3 or 4 values will also be provided.

## 2.7 Interim Analyses

No interim analysis is planned for this trial. A Data Safety Monitoring Board (DSMB) will meet periodically to review the safety and scientific conduct of the study. At a minimum, the DSMB is to review adverse events and safety laboratory assessments after the first six subjects complete Day 5 of treatment, and again after the first 12 subjects complete Day 5 of treatment.

#### 3. DATA HANDLING

## 3.1 Baseline and Study Visits

Study Day 1 will be the day of randomization.

The summary of hospitalization status will be based on the Study Day (derived relative to the day of randomization).

For the summary of inflammatory markers, Baseline will be the last assessment prior to dosing (SOC plus brequinar group) or last assessment on or prior to Study Day 1 (SOC group). Post-baseline timepoints will be based on the Study Day (derived relative to the day of randomization), where Day 15 includes a 4-day window (Study Day 11-19). If there are multiple results on the same day, the earliest result will be used.

For all other summaries, post-baseline timepoints will use the visit as recorded on the case report form, and Baseline will be the last non-missing value prior to randomization, including unscheduled assessments. Otherwise, unscheduled data will not be used in the analyses, but will be presented in the listings.

#### 3.2 Derived Data

#### **Prior and Concomitant Medication/Procedure**

A prior medication/procedure is any medication/procedure that started prior to date of randomization. A concomitant medication/procedure is any medication/procedure that either has a start date on or after date of randomization, or is ongoing on the date of randomization.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


#### **Hospitalization Status**

If a subject experiences multiple hospitalization status types on the given day, the worst status will be summarized on the day of interest.

#### **NEWS2 Score**

Chart 1: The NEWS scoring system

| Physiological parameter | 3 | 2 | 1 | Score<br>0 | 1 | 2 | 3 |
|---|---|---|---|---|---|---|---|
| Respiration rate<br>(per minute) | <b>≤</b> 8 | | 9–11 | 12-20 | | 21–24 | ≥25 |
| SpO <sub>2</sub> Scale 1 (%) | ≤91 | 92–93 | 94–95 | ≥96 | | | |
| SpO <sub>2</sub> Scale 2 (%) | <b>≤</b> 83 | 84–85 | 86–87 | 88–92<br>≥93 on air | 93–94 on<br>oxygen | 95–96 on<br>oxygen | ≥97 on<br>oxygen |
| Air or oxygen? | | Oxygen | | Air | | | |
| Systolic blood<br>pressure (mmHg) | ≤90 | 91–100 | 101–110 | 111–219 | | | ≥220 |
| Pulse (per minute) | ≤40 | | 41–50 | 51–90 | 91–110 | 111–130 | ≥131 |
| Consciousness | | | | Alert | | | CVPU |
| Temperature (°C) | ≤35.0 | | 35.1–36.0 | 36.1–38.0 | 38.1–39.0 | ≥39.1 | |

Use Chart 1 NEW2 scoring system to derive NEW2 score of each physiological parameter collected from case report forms. If hypercapnic respiratory failure, use SpO2 Scale 2; otherwise use SpO2 Scale 1. The total possible score ranges from 0 to 20. If any one of the NEWS2 parameters is not available on the study visit, the NEWS2 score will not be derived.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


#### **Normalization**

In order to summarize inflammatory marker results across the laboratories which have different normal ranges, normalization will be performed. The scale model will be applied for data transformation using the scale normalization formula:

$$S = X \times \frac{ULNs}{ULNx}$$

where X represents an assay value from the local laboratory, ULN<sub>x</sub> is the ULN from the laboratory, and ULN<sub>s</sub> is the upper limit of normal (ULN) from Site 02. Markers that are performed only at the central laboratory will not be normalized.

### 3.3 Missing Data and Data Conventions

No imputation is planned for missing data.

The follow conventions will be used for data handling:

- If SARS-Cov-2 is "not detected" in specimen, the test result will be set to 0 for analysis.
- For DHO and brequinar concentration levels, samples below the lower limit of quantitation (LLOQ) will be set to half of the LLOQ value for the summary tables (LLOQ of DHO is 5 ng/mL, LLOQ of concentration level is 5 mcg/mL).
- If a laboratory test result is reported as "< xxx" or "> xxx", the value of "xxx" will be used for analysis.
- If a medication or procedure has an incomplete start date, it is assumed to have started prior to randomization, unless the month and year are after randomization.
- If a medication or procedure is not checked as ongoing and has an incomplete stop date, it is assumed to have stopped after randomization, unless the month and year are prior to randomization.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


#### 4. CHANGES FROM THE PROTOCOL

Plasma viral load was listed in the protocol (Section 11.3) but will not be collected.

Nasopharyngeal viral culture was not listed in the protocol but was added to the central laboratory assessments.

The mITT population was not included in the protocol, but will be used for all analyses instead of the ITT population.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020 

## APPENDIX 1 CTCAE V4.03 GRADING FOR LABORATORY VALUES

| Lab Test | Lab Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| Albumin | G/DL | 3 to <lln< td=""><td>2 to &lt;3</td><td>&lt;2</td><td>Clinical Review Needed: Life- threatening consequences; urgent intervention indicated</td></lln<> | 2 to <3 | <2 | Clinical Review Needed: Life- threatening consequences; urgent intervention indicated |
| Alkaline<br>Phosphatase | U/L | >ULN to<br>2.5xULN | >2.5xULN<br>to 5xULN | >5xULN to 20xULN | >20xULN |
| Alanine<br>Amino<br>Transferase | U/L | >ULN to<br>3xULN | >3xULN to<br>5xULN | >5xULN to 20xULN | >20xULN |
| Aspartate<br>Amino<br>Transferase | U/L | >ULN to<br>2.5xULN | >2.5xULN<br>to 5xULN | >5xULN to 20xULN | >20xULN |
| Bilirubin<br>Total | MG/DL | >ULN to<br>1.5xULN | >1.5xULN<br>to 3xULN | >3xULN to 10xULN | >10xULN |
| Calcium | MG/DL | >ULN to 11.5 | >11.5 to 12.5 | >12.5 to 13.5 | >13.5 |
| Calcium | MG/DL | 8 to <lln< td=""><td>7 to &lt;8</td><td>6 to &lt;7</td><td>&lt;6</td></lln<> | 7 to <8 | 6 to <7 | <6 |
| Creatinine | MG/DL | >ULN to<br>1.5xULN | >1.5xULN to 3xULN | >3xULN to 6xULN | >6xULN |
| Glucose | MG/DL | >ULN to 160 | >160 to 250 | >250 to 500 | >500 |
| Glucose | MG/DL | 55 to <lln< td=""><td>40 to &lt;55</td><td>30 to &lt;40</td><td>&lt;30</td></lln<> | 40 to <55 | 30 to <40 | <30 |
| Potassium | MMOL/<br>L | >ULN to 5.5 | >5.5 to 6 | >6 to 7 | >7 |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020 

| Lab Test | Lab Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| Potassium | MMOL/<br>L | Clinical Review<br>Needed: Check<br>Grade 2 and<br>reassign if not<br>symptomatic<br>and no<br>intervention<br>indicated | 3 to <lln< td=""><td>2.5 to &lt;3</td><td>&lt;2.5</td></lln<> | 2.5 to <3 | <2.5 |
| Sodium | MMOL/<br>L | >ULN to 150 | >150 to 155 | >155 to 160 | >160 |
| Sodium | MMOL/<br>L | 130 to <lln< td=""><td>-</td><td>120 to &lt;130</td><td>&lt;120</td></lln<> | - | 120 to <130 | <120 |
| Lymphocytes,<br>Absolute | 10^3/UL | - | >4 to 20 | >20 | - |
| Lymphocytes,<br>Absolute | 10^3/UL | 0.8 to <lln< td=""><td>0.5 to &lt;0.8</td><td>0.2 to &lt;0.5</td><td>&lt;0.2</td></lln<> | 0.5 to <0.8 | 0.2 to <0.5 | <0.2 |
| Neutrophils,<br>Absolute | 10^3/UL | - | - | <1 | Clinical Review Needed: Life- threatening consequences; urgent intervention indicated |
| Neutrophils,<br>Absolute | 10^3/UL | 1.5 to <lln< td=""><td>1 to &lt;1.5</td><td>0.5 to &lt;1</td><td>&lt;0.5</td></lln<> | 1 to <1.5 | 0.5 to <1 | <0.5 |
| Hemoglobin | G/DL | >0 to 2 | >2 to 4 | >4 | |
| Hemoglobin | G/DL | >ULN to<br>ULN+2 | >ULN+2 to<br>ULN+4 | >ULN+4 | |
| Hemoglobin | G/DL | 10 to <lln< td=""><td>8 to &lt;10</td><td>&lt;8</td><td>Clinical Review Needed: Life- threatening consequences; urgent intervention indicated</td></lln<> | 8 to <10 | <8 | Clinical Review Needed: Life- threatening consequences; urgent intervention indicated |
| Platelet Count | 10^3/UL | 75 to <lln< td=""><td>50 to &lt;75</td><td>25 to &lt;50</td><td>&lt;25</td></lln<> | 50 to <75 | 25 to <50 | <25 |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 17-Dec-2020


| Lab Test | Lab Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| White Blood<br>Cell | 10^3/UL | - | - | >100 | Clinical Review Needed: Clinical manifestations of leucostasis; urgent intervention indicated |
| White Blood<br>Cell | 10^3/UL | 3 to <lln< td=""><td>2 to &lt;3</td><td>1 to &lt;2</td><td>&lt;1</td></lln<> | 2 to <3 | 1 to <2 | <1 |

Note: For these laboratory tests, Grade 0 is assigned if result does not meet above ranges.


Doc No.: TMP-BS-01 Rev No.: 4.0

# CLEAR CREEK BIO. INC. PROPOSED TABLES and LISTINGS PROTOCOL CCB-CRISIS-01

Version 1.0 17-Dec-2020

# CLEAR CREEK BIO. INC. PROPOSED TABLES and LISTINGS PROTOCOL CCB-CRISIS-01

Version 1.0 17-Dec-2020

## **Signature Page**

The proposed tables and listings have been reviewed and approved by the following personnel:

#### Prosoft Personnel

| 1 10301t 1 C1301IIIC1 | | | |
|---|---|---|---|
| Title | Printed Name | Signature | Date |
| Manager, | Daisy Chen | DocuSigned by: | 17-Dec-2020 |
| Statistics | | Daisy Chen | |
| Associate Vice | Diane Tipping | Signer Name: Daisy Chen | 17-Dec-2020 |
| President, Statistics | | Signing Reason: I have reviewed this d<br>Signing Time 17-Dec-2020 1:30:59 P | ocument<br>M PST |
| | | 2 1939 P. 1939 | |
| CCB Personnel | | Signing Reason: I approve this docume | MICT |
| Title | Printed Name | Signing Time: 17-Dec-2020 4:33:16 P Signature Dackisignators 5:64D0E959E82FB0235 | Date |
| Vice President, | Barbara Powers, PhD | Backstyred by 0400E939E021 B0233 | 17-Dec-2020 |
| Clinical Operations | | Barbara Powers | |
| | | Signer Name: Barbara Powers | |
| | | Signing Reason: I approve this documer Signing Time: 17-Dec-2020 1:40:07 PM | |
| | | 57DEAAD17C2240FEA72C57ABA124 | |

# CLEAR CREEK BIO. INC. PROPOSED TABLES and LISTINGS PROTOCOL CCB-CRISIS-01

## **TABLES**

| BOLD = SAMP | LE IS PROVIDED. |
|---|---|
| <b>Table 14.1.1</b> | Summary of Population by Site and Treatment |
| <b>Table 14.1.2</b> | Summary of Subject Disposition by Site and Treatment (Modified Intent- |
| | to-Treat Population) |
| <b>Table 14.1.3</b> | Summary of Demographics and Baseline Characteristics by Treatment |
| | (Modified Intent-to-Treat Population) |
| <b>Table 14.1.4</b> | Summary of Medical History by Treatment (Modified Intent-to-Treat |
| | Population) |
| <b>Table 14.1.5.1</b> | Summary of Prior Medications by Treatment (Modified Intent-to-Treat |
| 10010 1001001 | Population) |
| Table 14.1.5.2 | Summary of Concomitant Medications by Treatment (Modified Intent-to- |
| 14010 1 1.1.5.2 | Treat Population) |
| Table 14.1.6.1 | Summary of Prior Procedures by Treatment (Modified Intent-to-Treat |
| 14010 14.1.0.1 | Population) |
| Table 14.1.6.2 | Summary of Concomitant Procedures by Treatment (Modified Intent-to-Treat |
| 14010 14.1.0.2 | Population) |
| <b>Table 14.2.1</b> | Summary of Hospitalization Status and Mortality Rate by Treatment and |
| 1 apre 14.2.1 | Visit (Modified Intent-to-Treat Population) |
| Table 14 2 2 1 | |
| <b>Table 14.2.2.1</b> | Summary of Kaplan Meier Estimates for Duration of Hospitalization by |
| E | Treatment (Modified Intent-to-Treat Population) |
| <b>Figure 14.2.2.2</b> | Duration of Hospitalization by Treatment (Modified Intent-to-Treat |
| T 11 14001 | Population) |
| <b>Table 14.2.3.1</b> | Summary of Kaplan Meier Estimates for Time to Death by Treatment |
| T1 44000 | (Modified Intent-to-Treat Population) |
| <b>Figure 14.2.3.2</b> | Time to Death by Treatment (Modified Intent-to-Treat Population) |
| <b>Table 14.2.4.1</b> | Summary of NEWS2 Scores by Treatment and Visit (Modified Intent-to- |
| | Treat Population) |
| <b>Table 14.2.4.2</b> | Summary of NEWS2 Parameters by Treatment and Visit (Modified |
| | Intent-to-Treat Population) |
| <b>Table 14.2.5</b> | Summary of Change from Baseline in SARS-CoV-2 Viral Load |
| | (copies/mL) by Treatment and Visit (Modified Intent-to-Treat |
| | Population) |
| <b>Table 14.2.6</b> | Summary of Change from Baseline in Inflammatory Markers by |
| | Treatment and Visit (Modified Intent-to-Treat Population) |
| <b>Table 14.2.7</b> | Summary of Change from Baseline in DHO Level (ng/mL) by Treatment |
| | and Visit (Modified Intent-to-Treat Population) |

| <b>Table 14.2.8</b> | Summary of Change from Baseline in Brequinar Concentration Level |
|---|---|
| | (mcg/mL) by Treatment and Visit (Modified Intent-to-Treat Population) |
| <b>Table 14.3.1.1</b> | Overall Summary of Treatment-Emergent Adverse Events by Treatment |
| | (Modified Intent-to-Treat Population) |
| <b>Table 14.3.1.2</b> | Summary of Treatment-Emergent Adverse Events by Treatment |
| | (Modified Intent-to-Treat Population) |
| Table 14.3.1.3 | Summary of Related Treatment-Emergent Adverse Events by Treatment |
| | (Modified Intent-to-Treat Population) |
| Table 14.3.1.4 | Summary of Serious Treatment-Emergent Adverse Events by Treatment |
| | (Modified Intent-to-Treat Population) |
| Table 14.3.1.5 | Summary of Treatment-Emergent Adverse Events Leading to Study |
| | Discontinuation by Treatment (Modified Intent-to-Treat Population) |
| Table 14.3.1.6 | Summary of Treatment-Emergent Adverse Events of Interest by Treatment |
| | (Modified Intent-to-Treat Population) |
| <b>Table 14.3.1.7</b> | Summary of Treatment-Emergent Adverse Events by Severity and |
| | Treatment (Modified Intent-to-Treat Population) |
| <b>Table 14.3.2</b> | Summary of Change from Baseline in Laboratory Parameters of Special |
| | Interest by Treatment and Visit (Modified Intent-to-Treat Population) |

## LISTINGS

| <b>Listing 16.2.1</b> | Listing of End of Study Status by Treatment |
|---|---|
| <b>Listing 16.2.2</b> | Listing of Inclusion/Exclusion Criteria and Randomization |
| <b>Listing 16.2.3</b> | Listing of Informed Consent and Study Populations by Treatment |
| <b>Listing 16.2.4.1</b> | Listing of Subject Demographics by Treatment |
| <b>Listing 16.2.4.2</b> | Listing of Medical History by Treatment |
| <b>Listing 16.2.4.3</b> | Listing of Prior and Concomitant Medications by Treatment |
| <b>Listing 16.2.4.4</b> | Listing of Prior and Concomitant Procedures by Treatment |
| <b>Listing 16.2.5.1</b> | Listing of Dosing Information (SOC + Brequinar Only) |
| <b>Listing 16.2.5.2</b> | Listing of PK/DHO Results by Treatment |
| <b>Listing 16.2.6.1</b> | Listing of NEWS2 Assessments by Treatment |
| <b>Listing 16.2.6.2</b> | Listing of Inflammatory Markers by Treatment |
| <b>Listing 16.2.6.3</b> | Listing of SARS-CoV-2 Viral Load and Viral Culture by Treatment |
| <b>Listing 16.2.6.4</b> | Listing of Hospitalization Log by Treatment |
| <b>Listing 16.2.6.5</b> | Listing of Survival Status by Treatment |
| <b>Listing 16.2.7.1</b> | Listing of Adverse Events by Treatment |
| Listing 16.2.7.2 | Listing of Related Adverse Events by Treatment |
| Listing 16.2.7.3 | Listing of Serious Adverse Events by Treatment |
| Listing 16.2.7.4 | Listing of Grade 3 or 4 Adverse Events by Treatment |
| <b>Listing 16.2.8.1.1</b> | Listing of Chemistry Laboratory Tests by Treatment |
| Listing 16.2.8.1.2 | Listing of Grade 3 or 4 Chemistry Laboratory Tests by Parameter and |
| | Treatment |
| Listing 16.2.8.2.1 | Listing of Hematology Laboratory Tests by Treatment |
| Listing 16.2.8.2.2 | Listing of Grade 3 or 4 Hematology Laboratory Tests by Parameter and |
| - | Treatment |
| Listing 16.2.8.3 | Listing of Urinalysis Laboratory Tests by Treatment |

#### **Conventions:**

- For categorical data:
  - Percents are displayed with one decimal
  - When displaying counts and percents, the percent is contained within parentheses and does not include the "%" symbol
  - If the count is zero, no percent is displayed
  - If missing data occurs, a "Missing" row will be added to the summary table. The count of missing will be presented (no percent). The percentages for remaining rows will be based on the number of non-missing responses (i.e., the denominator does not include the missing counts)
- For continuous data, rounding will be based on the following conventions unless otherwise specified
  - Min and Max displayed to the same number of decimals as the original data
  - Mean, Median, and other percentiles displayed to 1 more decimal than the original data
  - SE and CIs displayed to 2 more decimals than the original data

#### Summary of Populations by Site and Treatment

| | SOC + Brequinar<br>n (%) | SOC<br>n (%) |
|---|---|---|
| Overall | | |
| Randomized | xx | xx |
| Modified Intent-to-Treat <sup>a</sup> | xx (xx.x) | xx (xx.x) |
| Site xx | | |
| Randomized | XX | xx |
| Modified Intent-to-Treat <sup>a</sup> | xx (xx.x) | xx (xx.x) |

a: Modified Intent-to-Treat (mITT) population includes all randomized subjects who had at least one post-randomization assessment, and who received at least one dose of study medication if randomized to SOC + Brequinar group. Source: Listing 16.X.X.X

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.1.2 Summary of Subject Disposition by Site and Treatment Modified Intent-to-Treat Population

| | SOC + Brequinar | SOC |
|--------------------------------------|-----------------|-----------|
| | (N=xx) | (N=xx) |
| | n (%) | n (%) |
| Overall | | |
| Completed the study (through Day 15) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) |
| Physician Decision | xx (xx.x) | xx (xx.x) |
| Adverse Event | xx (xx.x) | xx (xx.x) |
| Withdrawal by Subject | xx (xx.x) | xx (xx.x) |
| Study Terminated by Sponsor | xx (xx.x) | xx (xx.x) |
| Protocol Violation | xx (xx.x) | xx (xx.x) |
| Lost to Follow-Up | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) |
| Site xx | | |
| Completed the study (through Day 15) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) |
| Physician Decision | xx (xx.x) | xx (xx.x) |
| Adverse Event | xx (xx.x) | xx (xx.x) |
| Withdrawal by Subject | xx (xx.x) | xx (xx.x) |
| Study Terminated by Sponsor | xx (xx.x) | xx (xx.x) |
| Protocol Violation | xx (xx.x) | xx (xx.x) |
| Lost to Follow-Up | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) |
| Source: Listing 16.X.X.X | | |

Programming note: Sort in descending frequency based on the number of subjects in the SOC + Brequinar group, except for "Other" that shall stay at the last row. Sort alphabetically to break ties.

## Summary of Demographics and Baseline Characteristics by Treatment Modified Intent-to-Treat Population

| Parameter | SOC + Brequinar | SOC |
|-------------------------------------------|-----------------|--------------|
| | (N=xx) | (N=xx) |
| Age (years) | | |
| n | xx | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx |
| Sex, [n (%)] | | |
| Male | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) |
| Ethnicity, [n (%)] | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) |
| Race, [n (%)] | | |
| White | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) |
| Height (cm) | | |
| n | xx | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x(xx.xx) |
| Median | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX |
| Weight (kg) | | |
| n | xx | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x(xx.xx) |
| Median | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | XX.X, XX.X |
| Min, Max | xx, xx | XX, XX |
| BSA (m2) | | |
| n | xx | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx |
| Source: Listing 16.X.X.X | | |

## Summary of Demographics and Baseline Characteristics by Treatment Intent-to-Treat Population

| Parameter | SOC + Brequinar | SOC |
|---------------------------------------------|-----------------|--------------|
| | (N=xx) | (N=xx) |
| NEWS2 Score | | |
| n | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | xx, xx | xx, xx |
| ICU Level of Care at Randomization, [n (%)] | | |
| Yes | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) |
| Source: Listing 16.X.X.X | | |

### Summary of Medical History by Treatment Modified Intent-to-Treat Population

| System Organ Class<br>Preferred Term | SOC+ Brequinar<br>(N=xx) | SOC<br>(N=xx) |
|---|---|---|
| | n (%) | n (%) |
| Any Medical History Event | | |
| Overall | xx (xx.x) | xx (xx.x) |
| SOC 1 | | |
| Overall | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) |
| SOC 2 | | |
| Overall | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) |
| etc. | | |
| Note: Subjects reporting multiple occurrences of | f the same preferred term are only counted once | e within a given cell. |
| Source: Listing 16.X.X.X | | |

Programming note: Sort in descending frequency based on the number of subjects in the SOC+ Brequinar group. Sort alphabetically to break ties.

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.1.5.1 Summary of Prior Medications by Treatment Modified Intent-to-Treat Population

| Pharmacological Subgroup<br>Prior Medication | SOC+ Brequinar<br>(N=xx) | SOC<br>(N=xx) |
|---|---|---|
| | n (%) | n (%) |
| Any Prior Medication | | |
| Overall | xx (xx.x) | xx (xx.x) |
| Subgroup 1 | | |
| Overall | xx (xx.x) | xx (xx.x) |
| Medication 1 | xx (xx.x) | xx (xx.x) |
| Medication 2 | xx (xx.x) | xx (xx.x) |
| Subgroup 2 | | |
| Overall | xx (xx.x) | xx (xx.x) |
| Medication 1 | xx (xx.x) | xx (xx.x) |
| Medication 2 | xx (xx.x) | xx (xx.x) |
| etc. | | |
| Note: Subjects reporting multiple medications of | the same coded term are only counted once with | in a given cell. |
| Source: Listing 16.X.X.X | | |

Programming note: Sort medications in descending frequency based on the number of subjects in the SOC + Brequinar group. Sort alphabetically to break ties. Pharmacological Subgroup comes from ATC3. If ATC3 is not available, use ATC2

Change column header to "System Organ Class Preferred Term" for Procedure tables.

## Summary of Hospitalization Status and Mortality Rate by Treatment and Visit Modified Intent-to-Treat Population

| Study Day | SOC + Brequinar | SOC<br>(N-vv) |
|--------------------------|-----------------|-----------------|
| Hospitalization Status | (N=xx)<br>n (%) | (N=xx)<br>n (%) |
| Study Day 3 | II (70) | н (70) |
| Died | xx (xx.x) | xx (xx.x) |
| Hospitalized in ICU | xx (xx.x) | XX (XX.X) |
| Initial Hospitalization | xx (xx.x) | XX (XX.X) |
| Re-Hospitalization | xx (xx.x) | xx (xx.x) |
| Hospitalized (not ICU) | xx (xx.x) | XX (XX.X) |
| Initial Hospitalization | | · · · |
| • | xx (xx.x) | XX (XX.X) |
| Re-Hospitalization | xx (xx.x) | xx (xx.x) |
| Discharged | xx (xx.x) | xx (xx.x) |
| Initial Hospitalization | xx (xx.x) | xx (xx.x) |
| Re-Hospitalization | xx (xx.x) | xx (xx.x) |
| Missing | XX | XX |
| etc. | | |
| Study Day 15 | | |
| Died | xx (xx.x) | xx (xx.x) |
| Hospitalized in ICU | xx (xx.x) | xx (xx.x) |
| Initial Hospitalization | xx (xx.x) | xx (xx.x) |
| Re-Hospitalization | xx (xx.x) | xx (xx.x) |
| Hospitalized (not ICU) | xx (xx.x) | xx (xx.x) |
| Initial Hospitalization | xx (xx.x) | xx (xx.x) |
| Re-Hospitalization | xx (xx.x) | xx (xx.x) |
| Discharged | xx (xx.x) | xx (xx.x) |
| Initial Hospitalization | xx (xx.x) | xx (xx.x) |
| Re-Hospitalization | xx (xx.x) | xx (xx.x) |
| Missing | XX | XX |
| Day 29 Contact | | |
| Died | xx (xx.x) | xx (xx.x) |
| Alive | xx (xx.x) | xx (xx.x) |
| Missing | XX | xx |
| Source: Listing 16.x.x.x | 1 | |

Programming notes: summarize hospitalization status and death on Study Day 3, 5, 7, 15; summarize only death on Day 29. Include missing rows to capture unknown status.


PRAFT

YYYY-MM-DD

pgmid.sas

## Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.2.2.1

## Summary of Kaplan Meier Estimates for Duration of Hospitalization by Treatment

#### Modified Intent-to-Treat Population

| | SOC + Brequinar<br>(N=xx) | SOC<br>(N=xx) |
|---------------------------------|---------------------------|---------------|
| Total Patients Discharged | XX | XX |
| Number of Censored <sup>a</sup> | xx | XX |
| Not Discharged by Day 15 Visit | XX | XX |
| Did Not Complete Study | XX | XX |
| Q1 | xx | xx |
| Median | xx | xx |
| Q3 | xx | XX |

Note: Duration of hospitalization is defined as Study Day at time of initial discharge.

Source: Listing 16.x.x.x

a: Subjects who were not discharged by the Day 15 visit will be censored at the Day 15 visit. Subjects who did not complete the trial while still hospitalized will be censored at the date of last contact.


Prage 1 of 1

Prage 1 of 1

Prage 1 of 1

Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Figure 14.2.2.2 Duration of Hospitalization by Treatment Modified Intent-to-Treat Population

Note: Duration of hospitalization is defined as the Study Day at time of initial discharge. Subjects who were not discharged by the Day 15 visit will be censored at the Day 15 visit. Subjects who did not complete the trial while still hospitalized will be censored at the date of last contact.

Source: 16.x.x.x


PRAFT

YYYY-MM-DD

pgmid.sas

## Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.2.3.1

#### Summary of Kaplan Meier Estimates for Time to Death by Treatment

#### Modified Intent-to-Treat Population

| | SOC + Brequinar<br>(N=xx) | SOC<br>(N=xx) |
|---------------------------------|---------------------------|---------------|
| Number of Deaths | xx | xx |
| Number of Censored <sup>a</sup> | xx | xx |
| Alive at Day 29 Contact | xx | XX |
| Unknown | XX | XX |
| Q1 | xx | XX |
| Median | xx | xx |
| Q3 | XX | XX |

a: Subjects who are alive at the Day 29 contact will be censored at the Day 29 contact. Subjects whose Day 29 survival is unknown will be censored at the date of last contact.

Source: Listing 16.x.x.x


Prage 1 of 1

Prage 1 of 1

Prage 1 of 1

Clear Creek Bio., Inc.: Protocol CCB-CRISIS-01
Figure 14.2.3.2
Time to Death by Treatment
Intent-to-Treat Population

Note: Subjects who are alive at the Day 29 contact will be censored at the Day 29 contact. Subjects whose Day 29 survival is unknown will be censored at the date of last contact. Source: 16.x.x.x

## Summary of NEWS2 Scores by Treatment and Visit Modified Intent-to-Treat Population

| Visit | SOC + Brequinar<br>(N=xx) | | SOC<br>(N=xx) | |
|---|---|---|---|---|
| | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Baseline | <u> </u> | | | 1 |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | XX.X, XX.X | | xx.x, xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| 0-4 | xx (xx.x) | | xx (xx.x) | |
| 5-6 | xx (xx.x) | | xx (xx.x) | |
| 7 or Higher | xx (xx.x) | | xx (xx.x) | |
| Day 3 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| 0-4 | xx (xx.x) | | xx (xx.x) | |
| 5-6 | xx (xx.x) | | xx (xx.x) | |
| 7 or Higher | xx (xx.x) | | xx (xx.x) | |
| etc. | <u>.</u> | | | |
| Source: Listing 16.x.x.x | | | | |

Programming note: Include Day 3, 5, 7, 15.
## Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.2.4.2

### Summary of NEWS2 Parameters by Treatment and Visit

#### Modified Intent-to-Treat Population

| | | Brequinar<br>=xx) | | OC<br>=xx) |
|---|---|---|---|---|
| Parameter<br>Visit | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Systolic Blood Pressure (mm<br>Baseline | Hg) | | | |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| Day 3 | | | | |
| n | XX | XX | XX | xx |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| ••• | · | | | |
| Supplemental Oxygen<br>Baseline | | | | |
| Subject with value | XX | | XX | |
| Yes, [n (%)] | xx (xx.x) | | xx (xx.x) | |
| No, [n (%)] | xx (xx.x) | | xx (xx.x) | |
| | - | | | |
| Hypercapnic Respiratory Fai<br>Baseline | ilure | | | |
| Subject with value | XX | | XX | |
| Yes, [n (%)] | xx (xx.x) | | xx (xx.x) | |
| No, [n (%)] | xx (xx.x) | | xx (xx.x) | |
| Unknown, [n (%)] | xx (xx.x) | | xx (xx.x) | |
| etc. | | | | |
| Note: Percentages of Supplement the Subject with value. Source: Listing 16.x.x.x | ental Oxygen, Hypercapnic | Respiratory Failure and | Level of Consciousnes | ss Alert are based on |

Programming notes: summarize all NEWS2 parameters on Day 3, 5, 7, 15. CFB for Oxygen, Hypercapnic and Alert won't be provided.


PRAFT

YYYY-MM-DD

pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.2.5 Party of Change from Posseline in SAPS CoV 2 Viral Load (conjec/mL) h

# Summary of Change from Baseline in SARS-CoV-2 Viral Load (copies/mL) by Treatment and Visit Modified Intent-to-Treat Population

| | | Brequinar<br>=xx) | | OC<br>=xx) |
|---|---|---|---|---|
| Visit | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Baseline | , | · | | 1 |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | XX.X, XX.X | | xx.x, xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| Day 3 | · | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 5 | · | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| etc. | • | | | |
| Source: Listing 16.2.x | | | | |

Programming note: Include Day 3,5,7,15.

#### Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.2.6

# Summary of Change from Baseline in Inflammatory Markers by Treatment and Visit Modified Intent-to-Treat Population

| | | Brequinar<br>=xx) | SOC<br>(N=xx) | |
|---|---|---|---|---|
| Parameter<br>Visit | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Parameter 1 (unit), Norm | al Range=xx-xx | 1 | | 1 |
| Baseline | | | | |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | |
| Min, Max | XX, XX | | xx, xx | |
| Day 3 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 5 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| etc. | 1 | | | |
| Parameter 2 (unit), Norm<br>Baseline | al Range=xx-xx | | | |
| Source: Listing 16.x.x.x | | | | |

Programming note: Include all parameters from local and central labs on Day 3, 5, 7, 15.

#### Clear Creek Bio., Inc.: Protocol CCB-CRISIS-01 Table 14.2.7

# Summary of Change from Baseline in DHO Level (ng/mL) by Treatment and Visit Intent-to-Treat Population

| | | Brequinar<br>=xx) | SOC<br>(N=xx) | |
|---|---|---|---|---|
| Visit | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Baseline | | | | |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| Day 3 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 5 | · | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| etc. | , | | | |
| Source: Listing 16.x.x.x | | | | |

Programming note: Include Day 3, 5, 7, 15.

#### Clear Creek Bio., Inc.: Protocol CCB-CRISIS-01 Table 14.2.8

# Summary of Change from Baseline in Brequinar Concentration Level (mcg/mL) by Treatment and Visit

#### Intent-to-Treat Population

| | | Brequinar<br>=xx) | | OC<br>=xx) |
|---|---|---|---|---|
| Visit | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Baseline | | | | |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| Day 3 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 5 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 7 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Source: Listing 16.x.x.x | | | | |

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.3.1.1

### Overall Summary of Treatment-Emergent Adverse Events by Treatment Modified Intent-to-Treat Population

| | SOC + Brequinar<br>(N=xx)<br>n (%) | SOC<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|
| Subjects with 1 or more TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with 1 or more treatment-related TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with 1 or more Grade 3 or above TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with 1 or more TEAE leading to drug withdrawn | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with 1 or more TEAE leading to study discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with 1 or more serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with fatal TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with TEAE of interest | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total number of TEAEs | xx | XX | XX |
| Total number of study drug-related <sup>a</sup> TEAEs | xx | XX | XX |
| Total number of Grade 3 or above TEAEs | XX | XX | XX |
| Total number of TEAEs leading to drug withdrawn | XX | XX | XX |
| Total number of TEAEs leading to study discontinuation | XX | XX | XX |
| Total number of serious TEAEs | XX | XX | XX |
| Total number of TEAEs of interest | XX | XX | XX |
| a: Includes possible, probable and definite. Source: Listing 16.X.X.X | | | |

YYYY-MM-DD pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.3.1.2

# Summary of Treatment-Emergent Adverse Events by Treatment Modified Intent-to-Treat Population

| | SOC + Brequ | uinar (N=xx) | SOC (I | SOC(N=xx) | | N=xx) |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Subjects <sup>a</sup> n (%) | Events<br>n | Subjects <sup>a</sup><br>n (%) | Events<br>n | Subjects <sup>a</sup><br>n (%) | Events<br>n |
| Any Adverse Event | | | | | | |
| Overall | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| SOC 1 | | | | | | |
| Overall | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 3 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| SOC 1 | | | | | | |
| Overall | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred Term 3 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

a: Subjects experiencing one or more TEAEs are counted only once for each adverse event term.

Source: Listing 16.X.X.X

Programming note: Sort SOCs in descending frequency using total number of subjects in the SOC + Brequinar group, then sort preferred terms in descending frequency. Sort alphabetically to break ties.

YYYY-MM-DD pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Table 14.3.1.7

# Summary of Treatment-Emergent Adverse Events by Severity and Treatment Modified Intent-to-Treat Population

| | | S | OC + Brequ | iinar (N=xx) | ) | | SOC (N=xx) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Subjects <sup>a</sup><br>n (%) | Grade 1 <sup>b</sup> | Grade 2 <sup>b</sup> | Grade 3 <sup>b</sup> | Grade 4 <sup>b</sup> | Grade 5 <sup>b</sup><br>n | Subjects <sup>a</sup><br>n (%) | Grade 1 <sup>b</sup> | Grade 2 <sup>b</sup> | Grade 3 <sup>b</sup> | Grade 4 <sup>b</sup><br>n | Grade 5 <sup>b</sup> |
| Overall | | | | | | | | | | | | |
| Overall | xx (xx.x) | XX | XX | XX | XX | XX | xx (xx.x) | XX | XX | XX | XX | XX |
| SOC1 | · | | | | | | | | | | | |
| Preferred Term 1 | xx (xx.x) | XX | XX | XX | XX | XX | xx (xx.x) | XX | XX | XX | XX | XX |
| Preferred Term 2 | xx (xx.x) | xx | XX | XX | XX | XX | xx (xx.x) | XX | XX | XX | XX | XX |
| Preferred Term 3 | xx (xx.x) | XX | XX | XX | XX | XX | xx (xx.x) | XX | XX | XX | XX | XX |

a: Subjects experiencing one or more TEAEs are counted only once for each adverse event term.

Source: Listing 16.X.X.X

Programming note: Sort SOCs in descending frequency using total number of subjects in the SOC + Brequinar group, then sort preferred terms in descending frequency. Sort alphabetically to break ties.

b: Subjects experiencing one or more TEAEs are counted only once for each adverse event term and counted only by the maximum severity.

#### Clear Creek Bio., Inc.: Protocol CCB-CRISIS-01 Table 14.3.2

Summary of Change from Baseline in Laboratory Parameters of Special Interest by Treatment and Visit

Modified Intent-to-Treat Population

| | | Brequinar<br>=xx) | | OC<br>=xx) |
|---|---|---|---|---|
| Parameter<br>Visit | Visit | Change from<br>Baseline | Visit | Change from<br>Baseline |
| Parameter 1 (unit)<br>Baseline | , | | | |
| n | XX | | XX | |
| Mean (SE) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| Day 2 | · | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 3 | | | | |
| n | XX | XX | XX | XX |
| Mean (SE) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| etc. | | | | |
| Parameter 2 (unit)<br>Baseline | | | | |
| Source: Listing 16.x.x.x | | | | |

Programming note: Include selected lab parameters: AST, ALT, ALP, Total Bilirubin, Creatinine, Hemoglobin, WBC, Absolute Neutrophils, Absolute

YYYY-MM-DD pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.1

# Listing of End of Study Status by Treatment

| Site-Subject | Date of Last<br>Contact | Did the patient complete the study? | Primary Reason Did Not Complete | Comments |
|---|---|---|---|---|
| SOC + Brequinar | | | | |
| xx-xxxx | 9999-99-99 | Yes | | |
| xx-xxxx | 9999-99-99 | Yes | | xxxxxxxxxxxx |
| SOC | | | | |
| xx-xxxx | 9999-99-99 | No | xxxxxxxxxxx | xxxxxxxxxxxx |
| xx-xxxx | 9999-99-99 | Yes | | |

Page 1 of x YYYY-MM-DD **DRAFT** pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.2

#### Listing of Inclusion/Exclusion Criteria and Randomization

| Site-<br>Subject | Does the subject meet all<br>the Inclusion/Exclusion<br>criteria? | Criterion<br>Not Met | Comment / Explain Reason<br>for Ineligibility | Date of<br>Randomization | Time of Randomization | Treatment<br>Assignment | ICU Level of<br>Care at<br>Randomization |
|---|---|---|---|---|---|---|---|
| XX-XXXX | Yes | | | 9999-99-99 | 99:99 | SOC | No |
| XX-XXXX | No | Exclusion 2 | xxxxxxxxxx | | | | Yes |
| | | Inclusion 1 | xxxxxxxxxx | | | | |
| XX-XXXX | Yes | | | 9999-99-99 | 99:99 | SOC + Brequinar | No |
| XX-XXXX | No | Inclusion 3 | xxxxxxxxxx | | | | No |
| XX-XXXX | Yes | | | 9999-99-99 | 99:99 | SOC + Brequinar | Yes |
| XX-XXXX | Yes | | | 9999-99-99 | 99:99 | SOC | No |

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.3

#### Listing of Informed Consent and Study Populations by Treatment

| Site-Subject | Date of Informed Consent | Time of Informed Consent | Modified Intent-to-Treat Population <sup>a</sup> |
|---|---|---|---|
| SOC + Brequinar | | | |
| XX-XXXX | 9999-99 | 99:99 | Yes |
| XX-XXXX | 9999-99 | 99:99 | Yes |
| XX-XXXX | 9999-99 | 99:99 | Yes |
| SOC | | | |
| XX-XXXX | 9999-99 | 99:99 | xxx |
| xx-xxxx | 9999-99 | 99:99 | xxx |
| XX-XXXX | 9999-99 | 99:99 | XXX |

a: Modified Intent-to-Treat (mITT) population includes all randomized subjects who had at least one post-randomization assessment, and who received at least one dose of study medication if randomized to SOC + Brequinar group.

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.4.1 Listing of Subject Demographics by Treatment

| Site-Subject | Date of Birth | Age<br>(years) | Sex | Ethnicity | Race | Height (unit) | Weight (unit) | BSA<br>(m2) |
|---|---|---|---|---|---|---|---|---|
| SOC + Brequinar | | | | | | | | |
| xx-xxxx | 9999-99-99 | XX | Male | xxxxxxxxxxx | xxxxxxxxxxx | xxx (in) | xxx (lb) | X.X |
| xx-xxxx | 9999-99-99 | XX | Female | xxxxxxxxxxx | xxxxxxxxxxx | xxx (cm) | Not Done | |
| xx-xxxx | 9999-99-99 | XX | Male | xxxxxxxxxxx | Other: xxxxxxxxxxxx | Not Done | xxx (kg) | |
| SOC | | | | | | | | |
| xx-xxxx | 9999-99-99 | XX | XXXXX | xxxxxxxxxxx | xxxxxxxxxxx | XXXX | XXXX | X.X |
| xx-xxxx | 9999-99-99 | XX | xxxxx | xxxxxxxxxxx | xxxxxxxxxxx | XXXX | XXXX | X.X |
| xx-xxxx | 9999-99-99 | XX | xxxxx | xxxxxxxxxxx | Other: xxxxxxxxxxxx | XXXX | XXXX | X.X |

YYYY-MM-DD pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.4.2

#### Listing of Medical History by Treatment

| Site-Subject | Diagnosis and/or Procedure | System Organ Class / Preferred Term | Onset Date | <b>Resolution Date</b> |
|---|---|---|---|---|
| | | | | (Ongoing) |
| SOC + Brequ | inar | | | |
| xx-xxxx | COVD-19 | xxxxxxxxxx / xxxxxxxxxxx | 9999-99-99 | Ongoing |
| | xxxxxxxxx | xxxxxxxxxx / xxxxxxxxxxx | 9999-99-99 | 9999-99-99 |
| xx-xxxx | COVD-19 | | | |
| SOC | | | | |
| xx-xxxx | COVD-19 | xxxxxxxxxx / xxxxxxxxxxx | 9999-99-99 | Ongoing |
| | xxxxxxxxxx | xxxxxxxxxx / xxxxxxxxxxx | 9999-99-99 | 9999-99-99 |
| | xxxxxxxxx | xxxxxxxxxx / xxxxxxxxxxx | 9999-99-99 | 9999-99-99 |
| xx-xxxx | COVD-19 | xxxxxxxxxx / xxxxxxxxxxx | 9999-99-99 | Ongoing |

YYYY-MM-DD pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.4.3

#### Listing of Prior and Concomitant Medications by Treatment

| Site-<br>Subject | M: Medication or Treatment <sup>a</sup> P: Pharmacological Subgroup C: Coded Term | Indication | Start Date | Stop Date<br>(Ongoing) | Dose | Unit | Route | Prior/<br>Con <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| SOC + Bre | equinar | | | | | | | |
| xx-xxxx | M: xxxxxxxxxx P: xxxxxxxxxx C: xxxxxxxxxx | xxxxxxx | 9999-99-99 | 9999-99-99 | xxx | XXX | xxxxx | Р |
| xx-xxxx | M: xxxxxxxxxxx P: xxxxxxxxxx C: xxxxxxxxxx | xxxxxxx | 9999-99-99 | Ongoing | xxx | XXX | Other: xxxxx | Р, С |
| | M: xxxxxxxxxx P: xxxxxxxxxx C: xxxxxxxxxx | xxxxxx | 9999-99-99 | 9999-99-99 | XXX | XXX | xxxxx | С |
| SOC | | | <u>.</u> | | | | | |
| xx-xxxx | None | | | | | | | |
| xx-xxxx | M: xxxxxxxxxxx P: xxxxxxxxxx C: xxxxxxxxxx | xxxxxx | 9999-99-99 | Ongoing | XXX | Other: xxx | xxxxx | С |

a: P=Prior medication, C=Concomitant medication. A prior medication is any medication that started prior to date of randomization. A concomitant medication is any medication that either has a start date on or after date of randomization, or is ongoing on the date of randomization.

Programming Note: Pharmacological Subgroup comes from ATC3. If ATC3 is not available, use ATC2.

YYYY-MM-DD pgmid.sas

### Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.4.4

#### Listing of Prior and Concomitant Procedures by Treatment

| Site-<br>Subject | P: Procedure<br>S: System Organ Class<br>T: Preferred Term | Indication | Start Date | Stop Date<br>(Ongoing) | Dose | Unit | Route | Prior/<br>Con <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| SOC + B | requinar | | | | | | | |
| XX-<br>XXXX | P: xxxxxxxxxxx<br>S: xxxxxxxxxxx<br>T: xxxxxxxxxxx | xxxxxx | 9999-99-99 | 9999-99-99 | xxx | xxx | xxxxx | P |
| XX-<br>XXXX | P: xxxxxxxxxxx<br>S: xxxxxxxxxx<br>T: xxxxxxxxxx | xxxxxx | 9999-99-99 | Ongoing | XXX | xxx | Other:<br>xxxxx | Р, С |
| | P: xxxxxxxxxxx<br>S: xxxxxxxxxxx<br>T: xxxxxxxxxxx | xxxxxx | 9999-99-99 | 9999-99-99 | xxx | xxx | xxxxx | С |
| SOC | | 1 | | | 1 | • | | |
| XX-<br>XXXX | None | | | | | | | |
| XX-<br>XXXX | P: xxxxxxxxxx<br>S: xxxxxxxxxx<br>T: xxxxxxxxxx | xxxxxx | 9999-99-99 | Ongoing | xxx | Other: xxx | xxxxx | С |

a: P=Prior procedure, C=Concomitant procedure. A prior procedure is any procedure that started prior to date of randomization. A concomitant procedure is any procedure that either has a start date on or after date of randomization, or is ongoing on the date of randomization.

Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.5.1

Listing of Dosing Information (SOC + Brequinar Only)

| | Day 1 | | Day 2 | | Day 3 | | Day 4 | | Day 5 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site-Subject | Date of Dosing | Time of Dosing | Date of Dosing | Time of Dosing | Date of Dosing | Time of Dosing | Date of Dosing | Time of<br>Dosing | Date of Dosing | Time of<br>Dosing |
| XX-XXXX | 9999-99-99 | 99:99 | Not Done | | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 |
| xx-xxxx | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 |
| xx-xxxx | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | Not Done | |
| xx-xxxx | Not Done | | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 | 9999-99-99 | 99:99 |

### Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.5.2

#### Listing of PK/DHO Results by Treatment

| Site-Subject | Visit | Not Done | Date Collected | Time Collected | PK Result (mcg/mL) <sup>a</sup> | DHO Result (ng/mL) <sup>a</sup> |
|---|---|---|---|---|---|---|
| SOC + Brequinar | · | | | | · | |
| xx-xxxx | Day 1 | | 9999-99-99 | 99:99 | XXX | xxxx |
| | Day 3 | | 9999-99-99 | 99:99 | xxx | xxxx |
| | Day 5 | Not Done | | | | |
| | Day 7 | | 9999-99-99 | 99:99 | xxx | xxxx |
| | Day 15 | | 9999-99-99 | 99:99 | XXX | xxxx |
| SOC | | | | · | | |
| xx-xxxx | Day 1 | | 9999-99-99 | 99:99 | BLOQ (<5) | xxxx |
| | Day 3 | | 9999-99-99 | 99:99 | XXX | xxxx |
| | Day 5 | | 9999-99-99 | 99:99 | XXX | xxxx |
| | Day 7 | | 9999-99-99 | 99:99 | XXX | BLOQ (<5) |
| | Day 15 | | 9999-99-99 | 99:99 | XXX | xxxx |
| a: BLOQ = Below | Limit of Quantific | cation (limit of quant | tification in parentheses) | ' | 1 | |

YYYY-MM-DD Pgmid.sas

### Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.6.1

#### Listing of NEWS2 Assessments by Treatment

| Site-<br>Subject | Visit | Date and Time<br>Collected | SBP <sup>a</sup><br>(mmHg) | DBP <sup>a</sup><br>(mmHg) | Pulse<br>(Beats/Min.) | Respiration<br>(Breath/<br>Min.) | SpO <sub>2</sub> /<br>SaO <sub>2</sub><br>(%) | Temp.<br>(Celsius) | Supplemental Oxygen? | Hypercapnic respiratory failure? | Alert? | NEWS<br>2 Score |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC + Br | equinar | | | | | | | | | | | |
| xx-xxxx | Day 1 | 9999-99-99T99:99 | xxx | xxx | ND | XXX | XXX | XX.X | Yes | Yes | Yes | XX |
| | Day 3 | 9999-99-99T99:99 | XXX | xxx | xxx | XXX | XXX | XX.X | Yes | No | No | XX |
| | Day 5 | 9999-99-99T99:99 | XXX | xxx | xxx | XXX | ND | XX.X | No | Yes | No | XX |
| | Day 7 | Not Done | | | | | | | | | | |
| | Day 15 | 9999-99-99T99:99 | XXX | XXX | XXX | XXX | XXX | XX.X | No | Unknown | Yes | XX |
| SOC | | 1 | | | | | | | I | | | |
| xx-xxxx | Day 1 | 9999-99-99T99:99 | xxx | xxx | XXX | ND | xxx | xx.x | xxx | XXX | xxx | XX |
| | Day 3 | 9999-99-99T99:99 | xxx | xxx | XXX | XXX | xxx | ND | XXX | XXX | xxx | XX |
| | Unsche duled | | | | | | | | | | | |
| | Day 5 | 9999-99-99T99:99 | XXX | xxx | xxx | XXX | XXX | xx.x | XXX | XXX | xxx | XX |
| | Day 7 | 9999-99-99T99:99 | ND | ND | XXX | XXX | XXX | xx.x | XXX | XXX | xxx | XX |
| | Day 15 | 9999-99-99T99:99 | xxx | xxx | XXX | | | xx.x | xxx | XXX | xxx | xx |

Note: ND=Not Done

a: SBP=Systolic Blood Pressure, DBP=Diastolic Blood Pressure.

YYYY-MM-DD Program.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.6.2

#### Listing of Inflammatory Markers by Treatment

| Parameter | Visit | Not Done | Laboratory | Date and Time<br>Collected | Result | Abnormal? | Reference Range |
|---|---|---|---|---|---|---|---|
| SOC + Brequinar | | | | | | | |
| Site-Subject= x | x-xxx | | | | | | |
| Parameter 1 (unit) | Day 1 | | Local | 9999-99-99T99:99 | XX.X | High | |
| | Day 3 | | Local | 9999-99-99T99:99 | XX.X | High | |
| | Day 5 | | Central | 9999-99-99T99:99 | XX.X | | |
| | Day 7 | Not Done | | | | | |
| | Day 15 | | Local | 9999-99-99T99:99 | XX.X | | |
| Parameter 2 (unit) | Day 1 | | Local | 9999-99-99T99:99 | XX.X | Abnormal | |
| | Day 3 | | Local | 9999-99-99T99:99 | XX.X | | |
| | Unscheduled | | Local | 9999-99-99T99:99 | XX.X | | |
| | Day 5 | | Local | 9999-99-99T99:99 | XX.X | | |
| | Day 7 | Not Done | | | | | |
| | Day 15 | | Local | 9999-99-99T99:99 | XX.X | | |
| SOC | | | | <u> </u> | | | |
| Site-Subject= x | x-xxx | | | | | | |
| Parameter 1 (unit) | Day 1 | | Central | 9999-99-99T99:99 | XX.X | | |
| | Day 3 | | Central | 9999-99-99T99:99 | XX.X | | |
| | Day 5 | | Central | 9999-99-99T99:99 | XX.X | | |
| | Day 7 | | Central | 9999-99-99T99:99 | XX.X | | |
| | Day 15 | | Central | 9999-99-99T99:99 | xx.x | | |

Programming note: Include all data collected in local and central labs, including the tests done in both labs or done multiple times.

#### Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.6.3

#### Listing of SARS-CoV-2 Viral Load and Viral Cultureunit by Treatment

| Site-Subject | Visit | Not Done | <b>Date Collected</b> | Time Collected | Viral Load (copies/mL) | Viral Culture (unit) |
|---|---|---|---|---|---|---|
| SOC + Brequir | ıar | | | | | |
| xx-xxxx | Day 1 | | 9999-99-99 | 99:99 | | |
| | Day 3 | | 9999-99-99 | 99:99 | | |
| | Day 5 | Not Done | | | | |
| | Day 7 | | 9999-99-99 | 99:99 | | |
| | Day 15 | | 9999-99-99 | 99:99 | | |
| SOC | | | | | | |
| xx-xxxx | Day 1 | | 9999-99-99 | 99:99 | | |
| | Day 3 | | 9999-99-99 | 99:99 | | |
| | Day 5 | | 9999-99-99 | 99:99 | | |
| | Day 7 | | 9999-99-99 | 99:99 | | |
| | Day 15 | | 9999-99-99 | 99:99 | | |

YYYY-MM-DD Pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.6.4

# Listing of Hospitalization Log by Treatment

| Site-Subject | Event Type | Event Date |
|-----------------|--------------------|------------|
| SOC + Brequinar | | |
| XX-XXXX | xxxxxxxxxxx | 9999-99 |
| XX-XXXX | xxxxxxxxxxx | 9999-99 |
| | Other: xxxxxxxxxxx | 9999-99 |
| | xxxxxxxxxxx | |
| SOC | | |
| xx-xxxx | None | |
| XX-XXXX | Other: xxxxxxxxxxx | 9999-99 |
| | xxxxxxxxxxx | |

YYYY-MM-DD Pgmid.sas

### Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.6.5

#### Listing of Survival Status by Treatment

| Site-Subject | Visit | <b>Date of Contact</b> | Survival Status | Date of Death | Not Done, Comment |
|---|---|---|---|---|---|
| SOC + Brequi | nar | | | | |
| xx-xxxx | Day 1 – Day 15 | | Alive | | |
| | Day 29 Contact | 9999-99-99 | Alive | | |
| xx-xxxx | Day 1 – Day 15 | | Patient Died | 9999-99-99 | |
| xx-xxxx | Day 1 – Day 15 | | Alive | | |
| | Day 29 Contact | | | | Not Done: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| SOC | | | | | |
| xx-xxxx | Day 1 – Day 15 | | Alive | | |
| | Day 29 Contact | 9999-99-99 | Patient Died | 9999-99-99 | |
| xx-xxxx | Day 1 – Day 15 | | Alive | | |
| | Day 29 Contact | 9999-99-99 | Alive | | |

YYYY-MM-DD pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.7.1

#### Listing of Adverse Events by Treatment

| Site-<br>Subject | Adverse Event Term/ System<br>Organ Class/ Preferred Term | Onset Date and<br>Time/ Resolution<br>Date and Time | Continuing? | Outcome <sup>a</sup> | Severity | Causality | Action Taken<br>with Study<br>Treatment | Action<br>Taken | Serious? |
|---|---|---|---|---|---|---|---|---|---|
| SOC + Br | requinar | | | | | | | | |
| xx-xxxx | xxxxxx/ xxxxxxx / xxxxxx* | 9999-99-99T99:99/<br>9999-99-99T99:99 | Continuous | RG | Grade 2 | Definite | Drug<br>Interrupted | None | No |
| xx-xxxx | xxxxxx/ xxxxxxx / xxxxxxx | 9999-99-99T99:99/<br>9999-99-99T99:99 | Intermittent | RD | Grade 4 | Probable | Drug<br>Withdrawn | Treatment<br>Prescribed | No |
| | xxxxxx/ xxxxxxx / xxxxxxx | 9999-99-99T99:99/<br>9999-99-99T99:99 | Continuous | RS | Grade 1 | Possible | Unknown | Discontinued<br>Study | No |
| SOC | | | | | | | | | |
| xx-xxxx | xxxxxx/ xxxxxxx / xxxxxxx | 9999-99-99T99:99/<br>9999-99-99T99:99 | Intermittent | NR | Grade 5 | Unlikely | Not Applicable | Treatment Prescribed, Discontinued Study | Yes |
| | xxxxxxx/ xxxxxxx / xxxxxxx | 9999-99-99T99:99/<br>9999-99-99T99:99 | Continuous | UN | Grade 3 | Unrelated | Dose Not<br>Changed | None | No |
| xx-xxxx | None | | | | | | | | |

<sup>\*</sup> Not Treatment-Emergent (onset date is prior to the day of randomization

a: FA=Fatal, NR=Not Recovered/Not Resolved, RD=Recovered/Resolved, RS=Recovered/Resolved with Sequelae, RG=Recovering/Resolving, UN=Unknown.

YYYY-MM-DD Pgmid.sas

# Clear Creek Bio, Inc.: Protocol CCB-CRISIS-01 Listing 16.2.8.1.1

# Listing of Chemistry Laboratory Tests by Treatment

| Parameter | Visit | Not Done | Date and Time<br>Collected | Lab Name | Result | Abnormal? | CTCAE<br>Grade <sup>a</sup> | Reference Range |
|---|---|---|---|---|---|---|---|---|
| SOC + Brequinar<br>Site-Subject= xx-xxxx | | | | | | | | |
| Parameter 1 (unit) | Day 1 | | 9999-99-99T99:99 | XXX | XX.X | High | 2 | XX.X-XX.X |
| | Day 2 | | 9999-99-99T99:99 | XXX | XX.X | High | 2 | XX.X-XX.X |
| | Day 3 | | 9999-99-99T99:99 | XXX | XX.X | High | 2 | XX.X-XX.X |
| | Day 4 | | 9999-99-99T99:99 | xxx | XX.X | | 0 | XX.X-XX.X |
| | Day 5 | | 9999-99-99T99:99 | XXX | XX.X | | 0 | XX.X-XX.X |
| | Day 6 | | 9999-99-99T99:99 | XXX | XX.X | | 0 | XX.X-XX.X |
| | Day 7 | | 9999-99-99T99:99 | Other: xxx | XX.X | | 0 | XX.X-XX.X |
| | Day 15 | | 9999-99-99T99:99 | Other: xxx | XX.X | | 0 | XX.X-XX.X |
| Parameter 2 (unit) | Day 1 | | 9999-99-99T99:99 | xxx | XX.X | Abnormal | | XX.X-XX.X |
| | Day | | 9999-99-99T99:99 | XXX | XX.X | | | XX.X-XX.X |
| SOC<br>Site-Subject= xx-xxxx | | | | | | | | |
| Parameter 1 (unit) | Day 1 | | 9999-99-99T99:99 | xxx | xx.x | | 0 | XX.X-XX.X |
| | Day 2 | | 9999-99-99T99:99 | xxx | xx.x | | 0 | XX.X-XX.X |
| | Day 3 | | 9999-99-99T99:99 | xxx | xx.x | | 0 | xx.x-xx.x |
| | Day 4 | | 9999-99-99T99:99 | xxx | xx.x | | 0 | XX.X-XX.X |
| | Day 5 | Not Done | | | | | 0 | |
| | Day 6 | | 9999-99-99T99:99 | xxx | xx.x | | 0 | XX.X-XX.X |
| | Day 7 | | 9999-99-99T99:99 | XXX | xx.x | Low | 1 | XX.X-XX.X |
| | Day 15 | | 9999-99-99T99:99 | Other: xxx | XX.X | Low | 1 | XX.X-XX.X |
| a: Grades were derived usin | g CTCAE criteria | where applicab | le. Grade 0 was assigned | for values that did | l not meet a CTCA | E criteria. | · | |



#### **Certificate Of Completion**

Envelope Id: EF97B78FA0BD4089A86DE8A58A8ED301

Subject: Please DocuSign: CCB-CRISIS-01 SAP v1.0 2020-12-17.docx, CCB-CRISIS-01 Mocks v1.0 2020-12-17.docx

Source Envelope:

Document Pages: 60 Signatures: 6 Envelope Originator:

Certificate Pages: 5 Initials: 0 Diane Tipping

AutoNav: Enabled 996 Old Eagle School Rd

Envelopeld Stamping: Disabled Suite 1106

Time Zone: (UTC-05:00) Eastern Time (US & Canada) Wayne, PA 19087

d.tipping@prosoftclinical.com IP Address: 100.19.112.47

Sent: 12/17/2020 4:28:47 PM

Viewed: 12/17/2020 4:29:53 PM

Signed: 12/17/2020 4:31:12 PM

Sent: 12/17/2020 4:31:15 PM

Viewed: 12/17/2020 4:32:21 PM

Signed: 12/17/2020 4:34:09 PM

Status: Completed

#### **Record Tracking**

Status: Original Holder: Diane Tipping Location: DocuSign

12/17/2020 4:25:00 PM d.tipping@prosoftclinical.com

#### Signer Events Signature Timestamp

Daisy Chen

Daisy Chen
D.Chen@prosoftclinical.com

Manager, Biostatistics Qiuxu (Daisy) Chen

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

2B3FFE95-115C-431E-B126-300C7C7DAC74

Using IP Address: 69.136.93.119

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I have reviewed this document
I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 5/22/2020 3:01:14 PM

ID: edc55d18-a3ea-4040-9c52-2ba801cd124a

Diane Tipping

d.tipping@prosoftclinical.com

VP Biostatistics Prosoft Clinical

Security Level: Email, Account Authentication

(Required)

Diana Tipping

Signature Adoption: Pre-selected Style

Signature ID:

92A2CD2F-7756-4D0E-959E-82FB02359B17

Using IP Address: 100.19.112.47

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document
I approve this document

#### Electronic Record and Signature Disclosure:

Not Offered via DocuSign

**Signer Events Signature Timestamp** Barbara Powers Sent: 12/17/2020 4:34:13 PM Barbara Powers bpowers@clearcreekbio.com Viewed: 12/17/2020 4:39:43 PM Security Level: Email, Account Authentication Signed: 12/17/2020 4:40:11 PM (Required) Signature Adoption: Pre-selected Style Signature ID: 57DEAAD1-7C22-40FE-A72C-57ABA124E827 Using IP Address: 173.44.85.49 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document I approve this document

Electronic Record and Signature Disclosure: Accepted: 12/17/2020 4:39:43 PM

ID: 602703f1-c8af-4241-a59c-3ddd3fb840e0

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 12/17/2020 4:28:47 PM<br>12/17/2020 4:39:43 PM<br>12/17/2020 4:40:11 PM<br>12/17/2020 4:40:11 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Prosoft Clinical (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Prosoft Clinical:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: t.sammartino@prosoftclinical.com

#### To advise Prosoft Clinical of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at t.sammartino@prosoftclinical.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Prosoft Clinical

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to t.sammartino@prosoftclinical.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Prosoft Clinical

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to t.sammartino@prosoftclinical.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process.

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Prosoft Clinical as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Prosoft Clinical during the course of your relationship with Prosoft Clinical.